CLINICAL TRIAL: NCT02330120
Title: Effects of Dexmedetomidine and Propofol on Pulmonary Mechanics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, mediha turktan, Cukurova University, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: intensive care
Record Dates: First submitted 2014-11-17; First posted 2015-01-01 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Abnormal Respiratory Airway Resistance
Keywords: peak airway pressure; airway resistance; sedation; intensive care
MeSH Terms: interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- propofol (Experimental): Propofol infusion 0.5-2 mg/kg/h for sedation in mechanically ventilated patients
  Interventions: Drug: propofol
- dexmedetomidine (Active Comparator): dexmedetomidine infusion 0.2-0.7 mcg/kg/h for sedation in mechanically ventilated patients
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: propofol
  Arms: propofol
Drug: dexmedetomidine
  Arms: dexmedetomidine

SUMMARY:
The aim of this study is to compare the effects of dexmedetomidine and propofol on pulmonary mechanics in intensive care patients.

DETAILED DESCRIPTION:
The aim of this study is to compare the effects propofol and dexmedetomidine on pulmonary mechanics. Sixty patients mechanically ventilated in intensive care unit are included in this study. Patients are divided into two random groups, Group P (propofol) and Group D (dexmedetomidine). Propofol infusion 0.5-2 mg/kg/h is given to Group P patients and dexmedetomidine infusion 0.2-0.7 mcg/kg/h is given to Group D patients for sedation. Initial blood gas analysis, airway resistance (cmH2O/L/sec), positive end-expiratory pressure (PEEP, cmH20), frequency (breath/min), tidal volume (mL/min), minute volume (mL), peak airway pressure (cmH20), compliance (mL/cmH20), endtidal CO2 (mmHg), SvO2 (%) values are recorded. This parameters are evaluated with Drager Evita 4 ventilator and recorded on 5th,15th,30th,45th ve 60th minutes . Sedation is observed using Riker and Ramsey Sedation-Agitation Scale. Compliance of patients to mechanical ventilation is observed and recorded.

The primary outcome measures are airway resistance and peak airway pressure. Secondary outcome measure is sedation score.

ELIGIBILITY:
Inclusion Criteria:

* The patients mechanically ventilated in intensive care unit

Exclusion Criteria:

* Patients with contraindications for using propofol and dexmedetomidine

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
airway resistance | 60 minutes
  airway resistans measured by Evita 4 ventilator flow sensor
peak airway pressure values | 60 minutes
  peak airway pressure values provide the methods used to Evita 4 ventilator flow sensor

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

REFERENCES:
- [Background] Fernandes FC, Ferreira HC, Cagido VR, Carvalho GM, Pereira LS, Faffe DS, Zin WA, Rocco PR. Effects of dexmedetomidine on respiratory mechanics and control of breathing in normal rats. Respir Physiol Neurobiol. 2006 Dec;154(3):342-50. doi: 10.1016/j.resp.2006.02.002. Epub 2006 Mar 9. PMID 16527548
- [Background] Bang SR, Lee SE, Ahn HJ, Kim JA, Shin BS, Roe HJ, Sim WS. Comparison of respiratory mechanics between sevoflurane and propofol-remifentanil anesthesia for laparoscopic colectomy. Korean J Anesthesiol. 2014 Feb;66(2):131-5. doi: 10.4097/kjae.2014.66.2.131. Epub 2014 Feb 28. PMID 24624271